CLINICAL TRIAL: NCT03818451
Title: Co-ultra PEALut Enhances Neuronal Recovery Following Moderate Traumatic Brain Injury
Acronym: GLIA13
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Alfredo Conti, Associate Professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLIA13_1
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Traumatic Brain Injury
Keywords: Moderate brain trauma; Glialia; Neuroinflammation; Neuroprotection
MeSH Terms: conditions — Brain Injuries, Traumatic; Neuroinflammatory Diseases | interventions — co-ultraPEALut

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): All patients are treated by standard treatments according to patterns of severity and in the light of different variables, mainly represented by the conditions of cerebral hemodynamics. These procedures can be summarized as follows:
  * Surgical evacuation of hemorrhagic masses and brain contusion
  * Medical management aimed to maintenance of euvolemia and adequate brain perfusion. Prevention of secondary complications of critical illness included: preventive treatment of venous thromboembolism (VTE) and seizures
  * Patient who undergo surgical treatment, will recieve also postoperative intensive care treatments including: position of the head high, lower values of end-tidal CO2, sedation with reduced metabolic consumption of O2, increase in plasma osmolarity by administration of mannitol in controlled doses or hypernatremia, therapeutic CSF drainage
- Study Group (Experimental): Standard treatment plus specific treatment. The investigational agent, the co-ultraPEALut, is administered orally twice daily (every 12 h) for 180 days in association with the specific therapy (e.g., antiplatelet agents, anticoagulants, antiepileptic drugs) commonly administered to these patients and/or with drugs prescribed for comorbidities (i.e. diabetes, arterial hypertension).
  Interventions: Dietary Supplement: Co-ultraPEALut (Glialia)

INTERVENTIONS:
Dietary Supplement: Co-ultraPEALut (Glialia) — Co-ultraPEALut is administered to moderate traumatic brain injured patients for 180 days
  Other Names: Glialia
  Arms: Study Group

SUMMARY:
Traumatic brain injury (TBI) typically provokes secondary injury mechanisms, including the dynamic interplay between the ischemic, inflammatory, and cytotoxic processes. Moreover, such an impact induces a substantial level of cell death and results in the degeneration of the dendrites, thereby leading to persistent motor, sensory, and cognitive dysfunction. Previous studies have shown that the adult-born immature granule neurons in the dentate gyrus are the most susceptible of all the cell types in the hippocampus to damage following a moderate TBI due to a controlled cortical impact (CCI) device. Currently, there is no efficient approach available for avoiding immature neuron death or degeneration following TBI. Hence, this study aimed to assess the neuro-regenerative properties of co-ultramicronized PEALut (Glialia®), which is composed of palmitoylethanolamide (PEA) and the flavonoid luteolin (Lut), in an in vivo model of TBI, as well as in patients affected by TBI.

DETAILED DESCRIPTION:
Study Setting All patients affected by moderate TBI (Glasgow Coma Score 9-13) admitted to the neurosurgical department of the University Hospital of Messina, Italy, will be screened for recruitment.

Ethics The institutional review board (IRB) approved the study. Written consent will be obtained from each patient or the closest family member prior to the start of the study.

Study Design A randomized controlled single-blind study to assess the effects of co-ultraPEALut (Glialia®) administration in TBI patients will be carried out. The study is set to recruit at least 30 patients.

Recruited patients are randomly allocated to one of the two branches of the study: standard TBI treatment + Glialia® (Study Group) and standard TBI treatment (Control Group) in a 1:1 ratio using precompiled randomization tables.

General treatment

All patients will undergo standard treatments according to patterns of severity and in the light of distinct variables, mainly represented by the conditions of cerebral hemodynamics. These procedures can be summarized as follows:

* Surgical evacuation of hemorrhagic masses and / or "debridement" of outbreaks brain contusion;
* Medical management aimed to maintenance of euvolemia and adequate brain perfusion. Goals were a systolic blood pressure >90 mmHg and a cerebral perfusion pressure >60 mmHg. Prevention of secondary complications of critical illness included: preventive therapy of venous thromboembolism (VTE) using low molecular weight heparin (LMWH) and seizures using levetiracetam prophylactically for the first seven days after injury;
* Patient who underwent surgical treatment, received also postoperative intensive care treatments including: position of the head high, lower values of end-tidal CO2, sedation with reduced metabolic consumption of O2, increase in plasma osmolarity by administration of mannitol in controlled doses or hypernatremia, therapeutic CSF drainage.

Specific Treatment The investigations agent, the co-ultraPEALut, will be administered orally twice daily (every 12 h) for 180 days in association with the specific therapy (e.g., antiplatelet agents, anticoagulants, antiepileptic drugs) commonly administered to these patients and/or with drugs prescribed for comorbidities (i.e. diabetes, arterial hypertension).

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injuries
* Moderate trauma
* Glasgow Coma Score 9-13
* Loss of consciousness lasting >1 min
* post-traumatic amnesia >20 minutes
* CT scan Marshall Scale class II-VI.

Exclusion Criteria:

* Spinal cord injuries
* Pre-existing neurological disorders affecting the brain and/or the spinal cord
* Severe hypertension
* Diabetes, and chronic renal disease
* Remarkable chronic cerebravasculopathy of the CT
* Severe cognitive deficit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive outcome assessed Mini Mental State Examination (MMSE) | All patients will undergo neurological and neuropsychological evaluations at baseline (T0), after 30 days (T30) and 6 months (T180)
  Impairment of cognitive abilities will be evaluated by the Mini Mental State Examination (MMSE) (Folstein et al., 1975) adjusted for educational level and age. This is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time that is within the scope of this research. The threshold value for normal performance is set to 24 points. The outcome measure will be represented by the absolute score and by the change between the score recorded after 180 days and the baseline value
Cognitive outcome assessed by the Brief Neuropsychological Cognitive Examination (BNCE) | All patients will undergo neurological and neuropsychological evaluations at baseline (T0), after 30 days (T30) and 6 months (T180)
  Brief Neuropsychological Cognitive Examination (BNCE) (Ball et al., 2009). This consists in 10 subtests composed of easily administered tasks, none requiring more than minimal reading skills.Total score indicating overall severity of impairment (expressed in percentage), subtest scores, and two aggregate scores for the simple and complex subtests are provided as percentage of the maximum score. The outcome measure will be represented by the absolute score and by the difference between the score recorded after 180 days and the baseline value
Depression outcome assessed by Beck Depression Inventory | Outcome measure will be assessed at 180 days (T180) after trauma
  Depression will be assessed by the Beck inventory depression scale.This is a 21-question multiple-choice (scored 0-3 each) self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Scores will be categorized as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression
  Depression score will be assessed at 180 days (T180) after trauma
Assessment of Independence by Barthel Index | Outcome measure will be assessed at 180 days (T180) after trauma
  Independence in activities of daily living and self-care will be assessed by the Barthel Index. This is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. Each domain is scored in one-point increments with a full score of 20 indicating functional independence. Independence will be assessed at 180 days (T180) after trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided